CLINICAL TRIAL: NCT04641520
Title: A Comparative Study on Shoulder Rotational Strength and Range of Motion Between Unilateral and Bilateral Overhead Elite Athletes
Brief Title: Shoulder Profile Among Swimmers and Badminton Players
Acronym: SPASB
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Principal Investigator, Joffrey DRIGNY, Chief resident, Sport medicine department, University Hospital, Caen
Other Study IDs: SPASB
Record Dates: First submitted 2020-11-18; First posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Sport Injury; Shoulder Injuries
MeSH Terms: conditions — Shoulder Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Shoulder clinical testing with isokinetic strength assessment — All the participants had a shoulder clinical testing including shoulder rotators range of motion and isokinetic rotator muscle strength testing

SUMMARY:
Background: To compare the pre-season clinical measures with shoulder rotator strength and range of motion between bilateral (swimmers) and unilateral (badminton players) overhead athletes. Design: Prospective cohort study Participants: 42 athletes were enrolled including 24 elite badminton players and 18 elite swimmers Independent variables: A pre-season visit consisted in clinical and isokinetic shoulder strength testing. Clinical testing consisted in the shoulder range of motion (ROM) measurements aIsokinetic internal and external rotator shoulder muscles strength was tested at 60. Conventional and functional (eccentric-to-concentric) ratios (FR) were calculated.

ELIGIBILITY:
Inclusion Criteria:

* All the elite badminton players from a high-level club and the National Institute of Sport, Expertise, and Performance
* All the elite swimmers a high-level club

Exclusion Criteria:

* Players who had SSI in the 3 months prior to the isokinetic test or had shoulder surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Elite swimmers and badminton players
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Baseline Isokinetic strength testing (peak torques) | one preseason evaluation (september 2017 or september 2018 or september 2019)
  Shoulder rotator muscles isokinetic strength test, Measures: Peak Torque on internal rotator muscles (IR) and external rotator muscles (ER), in NM (newton.meter)
Baseline Isokinetic strength testing (ratios) | one preseason evaluation (september 2017 or september 2018 or september 2019)
  Shoulder rotator muscles isokinetic strength test, Measures: ratios between external rotator muscles (ER) and internal rotator muscles (IR) (ER:IR), in percent (%)
Clinical measurements, ROM | one preseason evaluation (september 2017 or september 2018 or september 2019)
  Shoulder internal and external rotation range of motion (ROM)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen Normandie, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided